CLINICAL TRIAL: NCT02192268
Title: ASSESSMENT OF THE EFFECTIVENESS OF HIGH FREQUENCY ORAL OSCILLATION AND MASK OF PEP IN CHILDREN WITH PNEUMONIA
Brief Title: Assesment of the Effectiveness of High Frequency Oral Oscillation and Mask of PEP in Children With Pneumonia
Acronym: PEP/HFOO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: University of Nove de Julho (Other); Hospital e maternidade São Luiz (Unknown)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, PhD, PhD, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEP/HFOO
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HFOO (Active Comparator): Children of the HFOO group will be subjected to two daily sessions of this resource which should be the same throughout her hospitalization with Shaker equipment.
  Interventions: Other: HFOO
- Assisted Coughing (Active Comparator): The children in the control group will be subjected to two daily sessions of assisted coughing.
  Interventions: Other: Assisted Coughing
- PEP (Active Comparator): The children will be subjected to PEP group two daily sessions of this resource which should be the same throughout her hospitalization with facial mask and valve Spring load with expiratory pressure of 10cmH2O.
  Interventions: Other: PEP

INTERVENTIONS:
Other: PEP
  Arms: PEP
Other: HFOO
  Arms: HFOO
Other: Assisted Coughing
  Arms: Assisted Coughing

SUMMARY:
The hypothesis of this study is that the physiologic effects of these (PEP/ HFOO) resources may have positive effects in this population of children with acute respiratory illness.

Thinking about this physical and physiological issue and due to the absence of a study that has evaluated the effectiveness of these instruments in patients with pneumonia, the objective of this study is to evaluate the short-term effects OOAF and mask of EPAP in children hospitalized for community-acquired pneumonia.

DETAILED DESCRIPTION:
The pneumonia is characterized by an acute infectious and inflammatory process, usually compromises the alveoli, bronchioles and interstitial space difficulting hematosis and may be in some or all of the cells filled with liquid and blood cells. The accumulation of secretion occurs as a consequence of this infectious and inflammatory process and contributes to clinical worsening by increasing airway resistance.

Respiratory physiotherapy has been questioned in patients with pneumonia and recent clinical studies have shown that there is no benefit to these patients. Respiratory physical therapy in addition to manual techniques has in his repertoire instrumental resources such as therapeutic high-frequency oral oscillator (HFOO) and the mask of expiratory positive pressure (PEP). The hypothesis of this study is that physical and physiological effects of these resources may have positive effects in this population of children with acute respiratory illness. The aim of this study is to evaluate the short-term effects HFOO and mask of PEP in children hospitalized for community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* age between 03 and 11 years old;
* have Pneumonia diagnosis done by a physician pediatrician (1) presence of cough and/or fever; (2) tachypnea according to age group (1-5 years-40 bpm; 5 years -30 bpm); (3) radiological change with consolidation or infiltrators associated or not with other findings compatible with pneumonia. All films will be evaluated by a radiologist and a pediatrician

Exclusion Criteria:

* chronic neurological Disease, or respiratory arrest
* failure to collaborate with therapy or assessment
* need of invasive or non-invasive ventilatory assistance
* hemodynamic instability
* vomiting or nausea
* not drained Pneumothorax
* not drained extensive pleural effusion
* dyspnea
* do not agree with research

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-08-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in Severity Score | Change from Baseline Severity score at 4 days
  Will be assigned a severity score proposed based on other studies with clinical variables and diagnostic criteria. This score will vary from 0 to 18 points. Participants will be followed for the duration of hospital stay, an expected average of 4 or 5 days.

SECONDARY OUTCOMES:
Change in Peak Flow meter | Change from Baseline peak flow at 4 days
  Peak Flow will be held three measurements in standing position with nasal clip with MedicateTM equipment with ATS range (60 to 900lmin) adult and pediatric use. Participants will be followed for the duration of hospital stay, an expected average of 4 or 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Evelim FD Gomes, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Hospital são Luiz Jabaquara, São Paulo, São Paulo, Brazil